CLINICAL TRIAL: NCT04291534
Title: Quality of Life and Addiction Among Hospital Night Workers - Descriptive Study of APHP Workers in Paris
Brief Title: Quality of Life and Addiction Among Hospital Night Workers
Acronym: ALADDIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Paris 7 - Denis Diderot (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Principal Investigator, Dr Martin Duracinsky, Principal Investigator, University Paris 7 - Denis Diderot
Other Study IDs: ALADDIN-QoLHospWork
Record Dates: First submitted 2020-02-04; First posted 2020-03-02 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Health Services Research; Quality of Life; Addiction; Substance-Related Disorders; Health Personnel
MeSH Terms: conditions — Behavior, Addictive; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The current context of the Covid-19 health crisis leads to an over-solicitation of health systems, with hospital staff in the front line. These personnel are undergoing high levels of stress, an alteration of their life rhythm, but also of their health status and quality of life at work. In addition, night work, through the disruption of circadian rhythms, has consequences on physical and mental health. The more frequent worsening of the condition of certain patients at night increases the burden and responsibilities of night staff. Increasing the use of psychoactive substances (SPAs) can become a solution for managing stress, work rhythms, sleep disorders and their consequences. This self-medication behaviour is not without risks, neither for staff nor for patients.

The ALADDIN study is a project made up of 2 waves of questionnaires - one during and the other after the Covid "hospital" crisis - filled in by the hospital night staff of AP-HP. This project will assess the impact of the Covid-19 epidemic on the quality of work life, mental health disorders, post-traumatic stress and substance use of hospital night staff.

The main objectives of this study is to evaluate the prevalence of psychoactive substance consumption among the night shift healthcare workers of the AP-HP and to describe the participants' quality of working life.

Methods The study is prospective study using an online self-completed questionnaire. The questionnaire was elaborated on the basis of the validated scales ASSIST (Alcohol, Smoking, and Substance Involvement Screening Test), AUDIT-C (Alcohol Use Disorder Test, shortened version) and HAD (for anxiety and depression) and on qualitative interviews conducted among care staff working the night shift.

The questionnaire will be completed at t0 (baseline) and 18 months after. This study will provide data on the consumption psychoactive substances by night hospital workers adn their quality of working life. It will also allow us to compare their consumption with the general population, and to describe the risk factors influencing the consumption.

ELIGIBILITY:
Inclusion Criteria:

- hospital workers at APHP, working at night or night and day alternance (working at least 3 hours between 9 p.m and 6 a.m, 2 times a week)

Exclusion Criteria:

* Hospital workers working during the day
* Workers working less than 3 hours a night two time a week
* Doctors

Ages: 16 Years to 67 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: As night workers are more prone to impaired health and to addictions, the study focuses on hospital night workers who represent a population particularly at risk.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Substance use prevalence | at T0 month : baseline
  Prevalence in APHP health workers of psychoactive substance consumption during the Covid 19 outbreak
Quality of working life scale | at T0 month : baseline
  Evaluation of the quality of working life during the Covid 19 outbreak using a validated scale

SECONDARY OUTCOMES:
Intervention preference | at T0 month
  Identify the preferences for intervention to improve the quality of life or change the addictive risk of night hospital staff at the APHP. Preferences for intervention methods and ranking of the least preferred.
Psychoactive substance consumption and associated factors | at T0 month
  Describe the risk factors associated with the consumption of psychoactive substances (PAS).
  Logistic or fish linear regression depending on the type of variable taken into account.
Impact of substance consumption on quality of life at work | at T0 month
  Evaluate the impact of substance use on quality of life at work Principal component analysis and classification to see if there are consumer groups for the night and / or day population. Method for taking into account missing, unused or invalid data
Risk factors associated with tobacco use | at T0 month
  Describe the risk factors associated with tobacco use among night hospital workers,
Impact of sleep quality on quality of working life and perceived health | at T0 month
  Evaluate the impact of sleep quality on the quality of working life and perceived health of night staff
Impact of anxiety and depressive symptoms on sleep and QWL. | at T0 month
  Describe the links between QWL and sleep, anxiety, depressive syndromes, and workplace upheaval.
Impact of sleep and workplace upheaval on anxiety and depressives symptoms | at T month
  Describe the links between anxiety/depressive syndromes and workplace disruption, sleep, and the Covid epidemic.
Modification of quality of working life score and psychoactive substances consumption prevalences | T18 months
  Comparison between the baseline score and prevalences and the score and prevalences 18 months after
Comparison of modification of quality of life score and declared quality of life modification after 18 month | T18 months
  Analysis of the relation between declared change and evolution of the quality of life score

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital de Bicêtre, Le Kremlin-Bicêtre
  - Assistance Publique des Hopitaux de Paris, Paris